CLINICAL TRIAL: NCT04642183
Title: Evaluation of Repeated, In-Clinic, Self-Imaging by NV-AMD Patients Using the Notal Vision Home OCT
Brief Title: Single In-Clinic Encounter With the Notal Vision Home OCT
Status: Completed | Type: Observational
Sponsor: Notal Vision Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: C2020.005
Record Dates: First submitted 2020-11-11; First posted 2020-11-24 (Actual); Last update posted 2021-12-23 (Actual); Status verified 2021-06

CONDITIONS: Neovascular Age-related Macular Degeneration; Intermediate Age Related Macular Degeneration (Disorder)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
this is a single In-Clinic Encounter With the Notal Vision Home OCT study. The study population will include up to 50 Age-related Macular Degeneration patients diagnosed with wet NV-AMD in at least one eye at the time of enrollment. All enrolled subjects should have at least one eye with active (wet) CNV (SRF and/or IRF) at the time of enrollment. All subjects will be enrolled at 1 site in the United States. in this study patients will be placed in a room with the Notal Vision Home OCT device and following a completion of a self tutorial will perform 3 unsupervised self-scans on each study eye (with a rest of ~5 minutes between self-scans). at the end of the testing sessions, the subject will be asked to complete subject user questionnaire.

DETAILED DESCRIPTION:
Office Visit:

At the enrollment Office Visit, the exams will be conducted in the following order:

1. Patient will be informed concerning the study and sign the Informed Consent Form (ICF) prior to conduct of any study procedures
2. The following data will be collected for each study subject:

   1. Subject's DOB (if allowed) or age
   2. Gender
   3. Number and type of injections and last injection date
3. Refraction correction
4. Snellen BCVA on both eyes on the day of the visit.
5. Eligible eyes of the subject will be scanned, non-dilated, with a Zeiss Cirrus OCT device 3 times with one (1) acceptable volume scan of each eye being obtained.

Scanning pattern to be used:

a. Macular cube, 6X6mm, 128 B-scans per volume scan NOTE: Any planned treatment for NV-AMD should be administered after completion of all study-related scans.

6. Eyes of the subject that meet all screening criteria will be enrolled. NOTE: All enrolled subjects should have at least one eye with active CNV (i.e., with SRF and/or IRF) confirmed by commercial OCT scan(s) at the time of enrollment 7. The following data will be collected for the study eye(s):

1. Qualifying diagnosis for the study eye from the subject's medical record
2. From the subject's medical record, the presence of other ophthalmic conditions including but not limited to:

i. Cataract ii. Glaucoma iii. Dry Eye iv. Other macula findings, e.g., epi retinal membrane, macular hole, vitreo-macular traction (VMT) Following confirmation of subject eligibility, subject will be placed in a room with the NVHO device which has been set up by a clinic technician.

1. The clinic technician will register the subject using the touchscreen of the NVHO device.
2. The subject will perform a self-tutorial, without any help from the clinic's staff. The training flow begins with demonstration clips followed by a practice phase. The training flow will be followed by a self-scan that the system uses as a calibration session.

   Note: If an eye cannot calibrate during 3 separate attempts or fails to test 3 consecutive times, the subject will discontinue self-imaging in this eye. If there is a fellow eye also enrolled in the study, the fellow eye will continue.
3. Following completion of the training and calibration session, the clinic technician sets the device for testing flows. The subject will perform three (3) unsupervised self-scans on each study eye with a rest period of ~5 minutes between self-scans. In case of scan failures, the user will perform up to 3 additional attempts to complete the required 3 self-scans. The number of attempts will not exceed 3 times per study eye.
4. At the end of each self-scanning, and during the 5-minute resting period, image results will be automatically uploaded to Notal Health Cloud.

   NOTE: Support provided by the sponsor will be available to study subjects throughout the study including tutorial, calibration and scanning, if needed.
5. Once the subject completes the testing session in its entirety, the subject will be asked to complete a questionnaire about their experience as a user of the NVHO device and proposed naming options for the device.
6. Collect AEs, if applicable.
7. Exit the subjects from the study.
8. Self-scan data will be backed up on the NVHO device. Commercial Cirrus OCT data will be copied to an external drive and sent to a Notal repository. Study visit data and subject questionnaires responses will be entered into a Sponsor-provided CRF and sent to a Notal repository.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to speak, read and understand English.
2. Ability to understand and agree to contents of informed consent either in writing or verbally.
3. Eighteen (18) years of age or older at the time of Informed Consent.
4. AMD patients diagnosed with wet NV-AMD in at least one eye (ie, with SRF, and/or IRF).
5. Fellow eye with NV-AMD (with or without fluid) or intermediate AMD.
6. Best corrected Visual Acuity of 20/320 or better in eyes participating at the study.

Exclusion Criteria:

1. Subjects with dilated pupils.
2. Any other retinal disease requiring steroidal or anti-VEGF injections.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include up to fifty (50) AMD patients diagnosed with wet NV-AMD in at least one eye at the time of enrollment. All subjects will be enrolled at one (1) site in the United States. Patients must meet all inclusion / exclusion criteria. All enrolled subjects should have at least one eye with active (wet) CNV (SRF and/or IRF) at the time of enrollment.
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2020-11-16 (Actual); Primary Completion 2021-08-24 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects who completed self-scanning following a self-tutorial. | 5-10 minutes
  Percentage of subjects who were able to perform a full self-scanning and generate a retinal volume scan.
Percentage of eyes that performed 4 self-scans with the same fluid status | About 30 min - upon completion of the study visit
  Percentage of eyes that performed 4 self-scans, where their fluid status (fluid present/absent) is identical based both human reader and the Notal OCT Analyzer (NOA) artificial-intelligence (AI) module.
Agreement between the Cirrus OCT and the NVHO device in detecting fluid in the central 3x3mm of the macula. | About 30 min - upon completion of the study visit
Summary of subject questionnaire results. | 5-10 minutes
  For the multi-choice questions - the average score (1-5) for each question. For open questions - collect the user's feedback for future improvements of the device

CONTACTS AND LOCATIONS:
Overall Officials: Michael Elman, MD, Principal Investigator — Michael Elman, M.D. 9114 Philadelphia Rd #310 Baltimore, Maryland 21237
Locations (1):
- Elman Retina Group, PA, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided